CLINICAL TRIAL: NCT03616561
Title: Observational Study on Quality of Life and Ultrasonographic Assessment of Nail Psoriasis After Treatment With Apremilast (JUST Study)
Brief Title: Quality of Life and Ultrasonographic Assessment of Nail Psoriasis After Treatment With Apremilast (JUST Study)
Acronym: JUST
Status: Completed | Type: Observational
Sponsor: Hospital de Granollers (Other)
Collaborators: Hospital de Sant Joan Despí Moisès Broggi (Other)
Responsible Party: Sponsor
Other Study IDs: 20172005
Record Dates: First submitted 2018-04-12; First posted 2018-08-06 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Nail Psoriasis
Keywords: Nail psoriasis; apremilast; ultrasound
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Apremilast: The cohort will be recruited in Hospital General de Granollers and Hospital Moises Broggi
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Target nail ultrasound will be performed in patients on apremilast by two expert dermatologists and each one will determine the ecographic parameters described in the protocol. These variables would be measured in one target nail in each patient, the greatest and most severely affected, at the investigator's criterion. The same nail will be assessed in all visits of the study (baseline, weeks 4, 16, 24, 38 and 52) . The ultrasound study will be performed with the same device in both hospitals: Esaote's MyLab ultrasound with a 20 MHz transducer. Prior to the start of the study the investigators evaluated the ultrasonographic inter-intraobserver concordance.
  Other Names: Nail ultrasound

SUMMARY:
Prospective open label non-randomized study, using Apremilast according to the manufacturer's Summary of Product Characteristics for 52 weeks, in patients with moderate to severe plaque psoriasis and nail psoriasis The study will be carried out in two hospital centers with experience in the management of patients with psoriasis and in the use of ultrasound of the nail apparatus. Visits and ultrasound would be performed by prescribing doctors themselves in their outpatient offices. Prior to the start of the study, the two doctors of each center will conduct a study to see the intraobserver and interobserver agreement on the ecographic parameters. The medication would be dispensed and controlled in the centers themselves and self-administered by patients at home. Each visit includes a ultrasound assessment of a target nail and measures of different scales: NAPSI, NAPPA.

DETAILED DESCRIPTION:
Primary objective:

- Determine the percentage of patients with at least a 20% improvement over the baseline visit of the NAPPA-PBI scale in weeks 4, 16, 24, 38 and 52.

Secondary objectives:

* Determine the percentage of improvement with respect to the baseline visit of the NAPPA QoL and CLIN scale in weeks 4, 16, 24, 38 and 52
* Determine the percentage of patients, regarding baseline visit, who reach a NAPSI 50 and changes in the NAPSI scale, in weeks 4, 16, 24, 38 and 52
* Determine the percentage of improvement or change of the nail ultrasound variables with respect to the baseline visit in weeks 4, 16, 24, 38 and 52
* Explore the possible correlation between clinical (NAPSI / NAPPA-Clin) and ultrasound variables before and after treatment
* Determine the percentage of patients with sonographic signs of enthesopathy of the distal interphalangeal joint before and after treatment
* Determine differences in clinical and sonographic parameters before treatment in good responders (NAPSI 50) compared to non-responders

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old at the time of signing the IC
* Patients with the diagnosis of plaque psoriasis, moderate to severe, at least 6 months before recruitment, with nail involvement and without active psoriatic arthropathy
* Nail involvement with a minimum NAPSI of 12 for fingernails, and any NAPSI for toenails
* Patients naïve to biological treatments
* In pregnant women, pregnancy must be ruled out before treatment can be started and they must use an effective contraceptive method to prevent pregnancy during treatment

Exclusion Criteria:

* Other major or clinically uncontrolled diseases
* Pregnancy or breastfeeding
* History of allergy to any component of the study medication
* Positivity for HBV surface antigen at the screening visit
* Positivity for HCV serology at the screening visit
* Active tuberculosis or inadequately treated history of tuberculosis
* Significant abnormalities in electrocardiogram at the screening visit
* Clinically significant abnormalities of the X-ray chest at the screening visit
* History of HIV infection or other acquired or congenital immunodeficiencies
* Active abuse or history of substance abuse 6 months prior to the screening visit
* Bacterial infection that required oral or injectable antibiotics or important viral or fungal infections within 4 weeks prior to the screening visit
* Malignancy or history of malignancy (other than cured in situ cutaneous squamous cell carcinoma or basal cell carcinoma, or in situ cérvix carcinoma without evidence of recurrence in the last 5 years)
* Rebound or relapse of psoriasis in the 4 weeks prior to the screening visit
* Presence of other cutaneous diseases that could interfere in the clinical assessment of the study
* Use of topical treatments that include corticosteroids, salicylic acid, urea> 10% or calcipotriol in the 2 weeks prior to the screening visit
* Use of systemic treatments for psoriasis, including systemic corticosteroids and PUVA or UVB phototherapy, within 4 weeks prior to the screening visit
* Previous or current use of biological treatments
* Use of any investigational drug within 4 weeks prior to the screening visit
* Previous treatment with apremilast

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with moderate to severe psoriasis vulgaris and nail involvement and are candidates for treatment with apremilast according to the product's summary of characteristics Moderate-severe psoriasis will be considered according to the consensus document of the Spanish group of psoriasis from the Spanish Academy of Dermatology and Venereology (AEDV, 2009)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2020-05-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Questionnaire: NAPPA- PBI changes | first visit and week 4, 16, 24, 38 and 52
  Nail assessment in psoriasis and psoriatic arthritis (NAPPA) is a modular instrument for the assessment of clinical and patient-reported outcomes in nail psoriasis. NAPPA comprises three components: NAPPA-QOL measuring nail-specific quality of life, NAPPA-PBI reflecting patient-relevant needs and treatment benefits, NAPPA-CLIN recording objective nail status. NAPPA-PBI questionnaire is a 24-item questionnaire which assesses patient-defined needs before and patient-rated benefits after treatment. The answers are given in Likert scales from 0 to 4, and a global score is calculated based on the importance-weighted benefit items. The principle of PBI is an advanced mode of goal attainment scaling with standardized goal items. range from 0 to 96. Higher values represent a better outcome.

SECONDARY OUTCOMES:
Nail ultrasound: changes in nail plate, bed and matrix thickness | baseline (first visit) and week 4, 16, 24, 38 and 52
  change in nail ultrasound measures nail plate, bed and matrix thickness. Data will be displayed in millimeters. Higher values represent a worse outcome.
Questionnaire: NAPPA-QoL changes | baseline (first visit) and week 4, 16, 24,38 and 52
  NAPPA-QOL questionnaire is a 20-item nail specific quality of life questionnaire which assesses specific quality of life conditions in the past week. Answers are given in Likert scales from 0 to 4. Factor analysis revealed three scales named 'Signs' (nail status), 'Stigma' (nail impact: stigma and emotional status), and 'Everyday life' (nail impact: everyday life). For use in clinical trials, a global score including all items without weighting is used and mean values are determined. range from 0 to 80. Higher values represent a worse outcome
Questionnaire: NAPPA- Clinical changes | baseline (first visit) and week 4, 16, 24, 38 and 52
  NAPPA-CLIN score is a simplified version of the NAPSI which only assesses the least and the worst involved nail of both hands, or both feet, respectively. Thus, the NAPPA-CLIN scores for hands or feet range from 0 to 16 respectively. Higher values represent a worse outcome
fingernail and toenail NAPSI score changes | baseline (first visit) and week 4, 16, 24, 38 and 52
  Nail psoriasis severity index (NAPSI) is a nail psoriasis-specific score, which in its original version comprises the assessment of matrix and nail bed involvement in every finger and toe by 8 criteria for each nail (0-8 point scale for every nail) .The NAPSI score will be determined using all 10 fingernails and toenails, on a 0-80 point scale (respectively). Higher values represent a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Muñoz, PhD, Principal Investigator — Hospital General de Granollers
Locations (1):
- Hospital General de Granollers, Granollers, Barcelona, Spain